CLINICAL TRIAL: NCT04038645
Title: Evaluation of Photobiomodulation on Nasal Fractures: a Randomized, Controlled, Double-blind Clinical Study
Brief Title: Evaluation of Photobiomodulation on Nasal Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Researcher will no longer conduct the study
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, Clinical Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nasal fracture
Record Dates: First submitted 2019-07-25; First posted 2019-07-31 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2019-12

CONDITIONS: Nasal Fracture
Keywords: Nasal Fracture; Photobiomodulation; Laser; Edema
MeSH Terms: conditions — Edema | interventions — Lasers; Control Groups

STUDY DESIGN:
Intervention Model Description: 36 patients will be allocated in the experimental and control groups: G1 - Experimental Group (n = 18 Photobiomodulation PBM) - the treatment will be performed in a conventional manner and the patient will receive laser at low intensity.
  G2 - Control group (n = 18 -placebo of PBM) - treatment will be performed in a conventional manner and simulation of PBM treatment.
Who Masked: Participant, Investigator
Masking Description: Only the researcher responsible for conducting the treatments (who will open the envelopes of the randomization) will know which treatment is assigned to each patient. The identification of each group will be revealed only after statistical analysis of the data for all those involved in the study by this researcher. Therefore, the researcher responsible for data collection (evaluation of edema and all secondary variables), the microbiologist and the statistician will be blind regarding the treatments assigned to the groups. The patient will also be blinded to the type of treatment performed, since the treatment with PBM will be identical in both groups and the treatment with PBM will be simulated in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (laser) (Active Comparator): The patients (n=18) will receive infrared LEDs in 6 points (3 on the right side and 3 on the left side) using a mask developed for the research . The irradiations will be performed with red LED ( wavelength = 660 nm) with output power of 100 milliwatt (mW) . The LED light outputs will be positioned in direct contact with the skin. During application of the LED both patient and operator will wear goggles.
  The red diode laser will be used. The power of the device is 100 mW and the wavelength used was 660nm (± 10nm). The diameter of the fiber optic of the apparatus has 600 μm, therefore a spot (area) of 0.002826cm2. The energy delivered per point is 1 Joule. 10 seconds of application is required. As 6 points are irradiated, the total energy delivered is 6 Joules. The energy density is 354 J / cm2 and the power density would be 35.4 W / cm2. The points will be determined by the same operator, obeying the protocol.
  Interventions: Other: Experimental group (laser)
- Control group (Placebo) (Placebo Comparator): The patients (n=18) will receive the LED at the same points recommended for the experimental group, but will be off. So that the patient does not identify the sound of activation of the device (beep), it will be recorded, and connected at the time of the application of the laser. The questionnaire to assess the impact of treatment on quality of life will be applied at baseline and after 8 days (by the same evaluator), as well as the evaluation of serum CRP.
  Interventions: Other: Control group (Placebo)

INTERVENTIONS:
Other: Experimental group (laser) — The patients will receive infrared LEDs in 6 points using a mask developed for the research . The irradiations will be performed with red LED ( wavelength = 660 nm) with output power of 100 milliwatt. During application of the LED both patient and operator will wear goggles.
  The red diode laser will be used. The power of the device is 100 mW and the wavelength used was 660nm (± 10nm). The diameter of the fiber optic of the apparatus has 600 μm, therefore a spot (area) of 0.002826cm2. The energy delivered per point is 1 Joule. 10 seconds of application is required. As 6 points are irradiated, the total energy delivered is 6 Joules. The energy density is 354 J / cm2 and the power density would be 35.4 W / cm2. The points will be determined by the same operator, obeying the protocol.
  Arms: Experimental Group (laser)
Other: Control group (Placebo) — Patients will receive the LED at the same points recommended for the experimental group, but will be off. So that the patient does not identify the sound of activation of the device (beep), it will be recorded, and connected at the time of the application of the laser. The questionnaire to assess the impact of treatment on quality of life will be applied at baseline and after 8 days as well as the evaluation of serum CRP.
  Arms: Control group (Placebo)

SUMMARY:
Nasal fractures are one of the most incidental of facial traumas. Regression of nasal edema is necessary so that surgical reduction of the fracture can be performed. It is known that photobiomodulation (PBM) reduces pain, edema and modulates inflammation. Regression of edema in a shorter time may decrease hospitalization time, decreasing hospital costs. However, there are no well-designed clinical studies on this subject. Therefore, the objective of this study will be to evaluate if PBM is able to reduce edema in the region of fractured nasal bones prior to nasal reduction and nasal packing, in order to reduce the patient's ability to go through surgery. Thirty-six patients diagnosed with a (primary) nasal fracture admitted to the Mandaqui Hospital Complex whose trauma occurred in the last 48 hours will be randomly divided into: G1- (control) (n = 18). . G2-Light emitter diode (LED) group (n = 18) - The standard hospital treatment will be performed + LED nasal mask. The main variable will be the edema evaluated by the same researcher and with the same technique. Secondary variables will be pain (visual analogue scale - VAS), temperature, rescue medication count, serum C-reactive protein and systemic inflammatory cytokines. Afterwards, the LED or its placebo will also be applied. The questionnaire to assess the impact of treatment on quality of life will be applied at the baseline and after 8 days. Adverse effects will be recorded and reported. If the data is normal, they will be submitted to Student's t-test. The data will be presented by their means ± standard deviation (SD) and the value of p will be set at 0.05.

DETAILED DESCRIPTION:
Nasal fractures are one of the most incidental of facial traumas. Regression of nasal edema is necessary so that surgical reduction of the fracture can be performed. It is known that photobiomodulation (PBM) reduces pain, edema and modulates inflammation. Regression of edema in a shorter time may decrease hospitalization time, decreasing hospital costs. However, there are no well-designed clinical studies on this subject. Therefore, the objective of this study will be to evaluate if PBM is able to reduce edema in the region of fractured nasal bones prior to nasal reduction and nasal packing, in order to reduce the patient's ability to go through surgery. Thirty-six patients diagnosed with a (primary) nasal fracture admitted to the Mandaqui Hospital Complex whose trauma occurred in the last 48 hours will be randomly divided into: G1- (control) (n = 18). The control group will be submitted to the standard hospital treatment: standard drug therapy (50mg diclofenac sodium - 5 days, 8 / 8h orally and 500mg dipyrone - 5 days, 6 / 6h , orally). Tylex 30mg orally will be given as rescue medication. In this group there will be simulation of the use of the mask. G2- LED group (n = 18) - The standard hospital treatment will be performed + LED nasal mask (3 points on each side of the nose), λ = 830nm, radiant exposure of 9.7 Joules J / cm2 for 10 minutes. Treatment will be performed at patient admission (up to 24 hours after nasal trauma), and at intervals explained below, for approximately 08 days after hospital admission. The main variable will be the edema evaluated by the same researcher and with the same technique. Secondary variables will be pain (visual analogue scale - VAS), temperature, rescue medication count, serum C-reactive protein and systemic inflammatory cytokines (TNF-α, interleukin-1 (IL-1), IL-6, IL-8 and IL- nasal fossa and saliva. All evaluations will be performed at baseline (T0) up to 48 hours after trauma, aiming at equivalence in the inflammatory process, (T1) 96h after trauma and (T2) 192h after trauma. Afterwards, the LED or its placebo will also be applied. The questionnaire to assess the impact of treatment on quality of life will be applied at the baseline and after 8 days. Adverse effects will be recorded and reported. If the data is normal, they will be submitted to Student's t-test. The data will be presented by their means ± SD and the value of p will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants.
* With a maximum of 48 hours after nasal trauma.

Exclusion Criteria:

* Patients using anticoagulant medication or use of medication that is anti-inflammatory chronically .
* Patients who report a hypersensitivity reaction to any drug used in the research
* Patients with previous nasal fractures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Edema | Throughout study completion on average of one year
  It will be applied a grading system for evaluating eyelid edema: 0 point, none; 1 point, minimal; 2 points, extending on to the iris; 3 points, covering the iris; 4 points, massive edema with the eyelid swollen shut.

SECONDARY OUTCOMES:
pain assessed by Vas | Throughout study completion on average of one year
  The pain will be assessed by applying a VAS visual analogic scale, consisting of a 100-mm line numbered in centimeters, with two closed ends. One end is labeled "0" and the other "100", meaning no pain and terrible pain, respectively. Each patient will be instructed to mark a vertical line with the point that best matches the intensity of pain during the evaluation. Instructions on marking will always be given to the patient by the same operator
Oral health related quality of life (OHRQoL) assessed by ohip-14 | Throughout study completion on average of one year
  Oral health related quality of life: using Oral Health Impact Profile (OHIP-14)questionnaire we will assess the impact on HRQOL will be measured. This instrument consists of 14 items arranged in 7 factors: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. The answers are given in a 5-point Likert scale (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = always).
C-reactive protein (CRP) | Throughout study completion on average of one year
  After approximately 4 to 24 hours of trauma, CRP serum levels reach peaks up to 1000 times its initial concentration, although it is a nonspecific marker and is closely related to tissue necrosis and inflammatory processes. The collection of 10 ml of peripheral blood will be performed through a specific tube by the nurses of the Mandaqui Hospital Group. This analysis will be performed at baseline and on the last assessment day.
temperature | Throughout study completion on average of one year.
  Temperature will be measured locally and systemically. The local measurement was measured using a Safety 1st® digital thermometer (Safety 1st®, "No Touch Forehead", Columbus, USA) in the nasal dorsum, one centimeter below the glabella.
Nasal Obstruction | Throughout study completion on average of one year.
  Nasal Obstruction - To evaluate nose permeability the following methodology will be used, the patient will be asked to numerically choose their sense of obstruction on a scale from zero to ten, zero represents no obstruction of air passage and ten indicates total obstruction. During evaluations the patient will not be allowed to see previous ratings. The patient should point out two numbers indicating that the score will be at an intermediate value. The result will be the average of both values. The value obtained will be multiplied by 10, for ease of comparison.
Bruise | Throughout study completion on average of one year.
  Periorbital bruise will be assessed in each patient by assessing the upper and lower eyelids separately, using a 0 to 4-point scale, Kargi scale, 2003
Salivary cytokines TNF-α, interleukin-1 (IL-1), IL-6, IL-8 and IL-10 | Throughout study completion on average of one year.
  5 ml of saliva sample will be collected in 50 ml tubes. They will be aliquoted (1.2ml) into 2 sterile microtubes and the samples will be stored at -80 ºC until further analysis of cytokines TNF-α, interleukin-1 (IL-1), IL-6, IL-8 and IL-10 via ELISA.
nasal exudate cytokines TNF-α, interleukin-1 (IL-1), IL-6, IL-8 and IL-10 | Throughout study completion on average of one year.
  Exudate samples will be collected with a paper cone that will be placed in the nasal cavity until resistance is felt. The cones will be placed in one sterile microcentrifuge tube and stored at -80 Celsius degree (ºC) until further analysis of cytokines TNF-α, interleukin-1 (IL-1), IL-6, IL-8 and IL-10 via ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina RT Horliana, Phd, Principal Investigator — Nove de Julho University (Uninove)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kargi E, Hosnuter M, Babuccu O, Altunkaya H, Altinyazar C. Effect of steroids on edema, ecchymosis, and intraoperative bleeding in rhinoplasty. Ann Plast Surg. 2003 Dec;51(6):570-4. doi: 10.1097/01.sap.0000095652.35806.c5. PMID 14646651
- [Background] Oliveira Sierra S, Melo Deana A, Mesquita Ferrari RA, Maia Albarello P, Bussadori SK, Santos Fernandes KP. Effect of low-level laser therapy on the post-surgical inflammatory process after third molar removal: study protocol for a double-blind randomized controlled trial. Trials. 2013 Nov 6;14:373. doi: 10.1186/1745-6215-14-373. PMID 24195796